CLINICAL TRIAL: NCT01184625
Title: Physical Exercise as a Targeted Therapy in Patients With Chronic Rheumatic Muscle Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: professor Ingrid Lundberg, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Exercise
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Myositis
Keywords: Myositis; Physical exercise; Disability
MeSH Terms: conditions — Myositis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Physical Exercise
- No intervention (No Intervention): 12 weeks of stable physical exercise level.

INTERVENTIONS:
Other: Physical Exercise — 12 weeks of physical exercise.
  Arms: Exercise

SUMMARY:
The objectives of this study are to test if hypoxia in muscle tissue is an important factor contributing to clinical symptoms in chronic rheumatic muscle inflammation and to evaluate if a 12 week endurance exercise program will improve muscle tissue hypoxia and disability in patients with chronic rheumatic muscle inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic, stable polymyositis or dermatomyositis with diagnosis of definite or probable polymyositis or dermatomyositis (Bohan and Peter 1975)
* Age 18-80 years
* Duration since diagnosis > 6 months
* Exercising < once a week,
* Stable disease activity and medication for at least one month.

Ten healthy controls matched for age, gender and physical exercise level will be included.

-

Exclusion Criteria:

* Severe pulmonary fibrosis
* Heart or lung conditions that contraindicate vigorous exercise
* Severe osteoporosis
* Not being able to perform the exercise program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Hypoxia related metabolites. | At baseline before intervention.
Hypoxia related metabolites. | After 12 weeks of endurance exercise intervention/ non intervention.

SECONDARY OUTCOMES:
Muscle impairment. | At baseline before intervention.
Muscle impairment. | After 12 weeks of endurance exercise intervention/ non intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid E Lundberg, MD, PhD, Prof, Principal Investigator — Rheumatology Unit, Department of Medicine, in Solna, Karolinska Institutet
Locations (1):
- Rheumatology unit, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Boehler JF, Hogarth MW, Barberio MD, Novak JS, Ghimbovschi S, Brown KJ, Alemo Munters L, Loell I, Chen YW, Gordish-Dressman H, Alexanderson H, Lundberg IE, Nagaraju K. Effect of endurance exercise on microRNAs in myositis skeletal muscle-A randomized controlled study. PLoS One. 2017 Aug 22;12(8):e0183292. doi: 10.1371/journal.pone.0183292. eCollection 2017. PMID 28829792
- [Derived] Alemo Munters L, Dastmalchi M, Katz A, Esbjornsson M, Loell I, Hanna B, Liden M, Westerblad H, Lundberg IE, Alexanderson H. Improved exercise performance and increased aerobic capacity after endurance training of patients with stable polymyositis and dermatomyositis. Arthritis Res Ther. 2013 Aug 13;15(4):R83. doi: 10.1186/ar4263. PMID 23941324
- [Derived] Alemo Munters L, Dastmalchi M, Andgren V, Emilson C, Bergegard J, Regardt M, Johansson A, Orefelt Tholander I, Hanna B, Liden M, Esbjornsson M, Alexanderson H. Improvement in health and possible reduction in disease activity using endurance exercise in patients with established polymyositis and dermatomyositis: a multicenter randomized controlled trial with a 1-year open extension followup. Arthritis Care Res (Hoboken). 2013 Dec;65(12):1959-68. doi: 10.1002/acr.22068. PMID 23861241